CLINICAL TRIAL: NCT02081924
Title: The Physiological Changes in Reproductive Hormones During Sustained Administration of Kisspeptin in Humans.
Brief Title: Reproductive Hormones During Sustained Administration of Kisspeptin
Acronym: KisspeptPump
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13/LO/1807
Record Dates: First submitted 2014-02-26; First posted 2014-03-07 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fertility Disorders; Hypothalamic Dysfunction
Keywords: Infertility; Kisspeptin; Reproductive hormones
MeSH Terms: conditions — Hypothalamic Diseases; Infertility | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-blinded placebo-controlled study. Women will receive an 8-h SC infusion of kisspeptin-54 0·1, 0·3 or 1·0 nmol/kg/h or saline in the early follicular phase of 4 separate menstrual cycles. Luteinising Hormone (LH), Follicle stimulating hormone (FSH) and oestradiol will be measured every 10 min during the infusions.
Who Masked: Participant
Masking Description: The participant won't know whether they are receiving placebo or which dose of kisspeptin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kisspeptin 0.1 (Active Comparator): Participants will receive kisspeptin hormone at a dose rate of 0.1nmol/kg/hour via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  Interventions: Other: Kisspeptin 0.1
- Saline (Placebo Comparator): Participants will receive placebo (saline) via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  Interventions: Other: Saline
- Kisspeptin 0.3 (Active Comparator): Participants will receive kisspeptin hormone at a dose rate of 0.3nmol/kg/hour via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  Interventions: Other: Kisspeptin 0.3
- Kisspeptin 1.0 (Active Comparator): Participants will receive kisspeptin hormone at a dose rate of 1.0nmol/kg/hour via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  Interventions: Other: Kisspeptin 1.0

INTERVENTIONS:
Other: Kisspeptin 0.1 — Participants will receive kisspeptin hormone at a dose rate of 0.1nmol/kg/hour via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  LH, FSH and oestradiol will be measured on day 1 and 8, at 10minute intervals for 8 hours and on Days 3 and 5 they will have a single blood measurement of the same hormones.
  Arms: Kisspeptin 0.1
Other: Saline — Participants will receive placebo (saline) via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  LH, FSH and oestradiol will be measured on day 1 and 8, at 10minute intervals for 8 hours and on Days 3 and 5 they will have a single blood measurement of the same hormones.
  Arms: Saline
Other: Kisspeptin 0.3 — Participants will receive kisspeptin hormone at a dose rate of 0.3 nmol/kg/hour via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  LH, FSH and oestradiol will be measured on day 1 and 8, at 10minute intervals for 8 hours and on Days 3 and 5 they will have a single blood measurement of the same hormones.
  Arms: Kisspeptin 0.3
Other: Kisspeptin 1.0 — Participants will receive kisspeptin hormone at a dose rate of 1.0 nmol/kg/hour via a subcutaneous pump device for 8 days during the early follicular phase of their menstrual cycle.
  LH, FSH and oestradiol will be measured on day 1 and 8, at 10minute intervals for 8 hours and on Days 3 and 5 they will have a single blood measurement of the same hormones.
  Arms: Kisspeptin 1.0

SUMMARY:
We want to find out what happens to reproductive hormone levels; Luteinising Hormone (LH), Follicle Stimulating Hormone (FSH), testosterone and oestradiol when kisspeptin is administered to people for a period of 8 days each month, using either placebo (saline) or kisspeptin in doses of 0.1, 0.3 or 1.0 nmol/kg/hour.

DETAILED DESCRIPTION:
Participants will be invited to have an initial baseline study to look at the hormone levels at regular intervals over the course of a day (8hours).

Following this, on a different day, volunteers will have an infusion of kisspeptin, which will be administered by a small pump to deliver the hormone into subcutaneous tissue (fatty tissue just below the skin surface). On day 1 of the pump infusion there will be another day of regular blood sampling for 8 hours. After this the kisspeptin pump will continue and the participants will return to the research unit on day 3 for a review and a single blood test. On day 5 the participants will have a review, a blood test and the kisspeptin pump will be changed. Kisspeptin infusion will continue and on Day 8 the participant will return for another 8 hour study. At the end of this the kisspeptin pump will be removed.

The above will be repeated using either placebo (saline) or kisspeptin in doses of 0.1, 0.3 or 1.0 nmol/kg/hour during the early follicular phase of 4 separate menstrual cycles.

ELIGIBILITY:
Inclusion criteria:

* Aged 18-60 years old
* Ability to give informed consent
* Secondary hypogonadism (or healthy participant)

Exclusion criteria:

* anaemia
* medical problems such as severe heart, kidney or liver disease
* blood donation in the last three months or intention to donate blood within 3 months of the end of the study
* needle phobia
* Poor venous access
* Active psychiatric illness
* Severe allergies
* Impaired ability to provide full consent to take part in the study
* Current alcohol or illicit drug dependence
* Current pregnancy or breast feeding
* Plans to conceive within 3 months of starting the study (barrier contraception must be used during and for 3 months after the end of the study)
* Arthritis or any impairment of hand coordination which would preclude using a hormone pump

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2014-04-02 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Kisspeptin on hypothalamic reproductive function - LH levels | 3 months
  Luteinising hormone levels will be measured at various time-points to assess the effect of kisspeptin on hypothalamic reproductive function, whilst the participant receives a kisspeptin infusion

SECONDARY OUTCOMES:
Effect of Kisspeptin on hypothalamic reproductive function - FSH levels | 3 months
  FSH levels will be measured at various time-points to assess the effect of kisspeptin on hypothalamic reproductive function, whilst the participant receives a kisspeptin infusion
Effect of Kisspeptin on hypothalamic reproductive function - Oestradiol levels | 3 months
  Oestradiol levels will be measured at various time-points to assess the effect of kisspeptin on hypothalamic reproductive function, whilst the participant receives a kisspeptin infusion
Do participants with normal fertility respond differently to sustained administration of kisspeptin, compared to participants with reduced fertility? | 3 months
  Reproductive hormone levels (LH, FSH, oestradiol) will be measured at various timepoints, whilst the participant receives a kisspeptin infusion. The results of the two groups will then be compared with one another.

CONTACTS AND LOCATIONS:
Overall Officials: Waljit Dhillo, PhD, FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhillo WS, Chaudhri OB, Patterson M, Thompson EL, Murphy KG, Badman MK, McGowan BM, Amber V, Patel S, Ghatei MA, Bloom SR. Kisspeptin-54 stimulates the hypothalamic-pituitary gonadal axis in human males. J Clin Endocrinol Metab. 2005 Dec;90(12):6609-15. doi: 10.1210/jc.2005-1468. Epub 2005 Sep 20. PMID 16174713
- [Background] Dhillo WS, Chaudhri OB, Thompson EL, Murphy KG, Patterson M, Ramachandran R, Nijher GK, Amber V, Kokkinos A, Donaldson M, Ghatei MA, Bloom SR. Kisspeptin-54 stimulates gonadotropin release most potently during the preovulatory phase of the menstrual cycle in women. J Clin Endocrinol Metab. 2007 Oct;92(10):3958-66. doi: 10.1210/jc.2007-1116. Epub 2007 Jul 17. PMID 17635940
- [Background] Jayasena CN, Nijher GM, Chaudhri OB, Murphy KG, Ranger A, Lim A, Patel D, Mehta A, Todd C, Ramachandran R, Salem V, Stamp GW, Donaldson M, Ghatei MA, Bloom SR, Dhillo WS. Subcutaneous injection of kisspeptin-54 acutely stimulates gonadotropin secretion in women with hypothalamic amenorrhea, but chronic administration causes tachyphylaxis. J Clin Endocrinol Metab. 2009 Nov;94(11):4315-23. doi: 10.1210/jc.2009-0406. Epub 2009 Oct 9. PMID 19820030
- [Background] Jayasena CN, Nijher GM, Abbara A, Murphy KG, Lim A, Patel D, Mehta A, Todd C, Donaldson M, Trew GH, Ghatei MA, Bloom SR, Dhillo WS. Twice-weekly administration of kisspeptin-54 for 8 weeks stimulates release of reproductive hormones in women with hypothalamic amenorrhea. Clin Pharmacol Ther. 2010 Dec;88(6):840-7. doi: 10.1038/clpt.2010.204. Epub 2010 Oct 27. PMID 20980998
- [Background] Jayasena CN, Nijher GM, Comninos AN, Abbara A, Januszewki A, Vaal ML, Sriskandarajah L, Murphy KG, Farzad Z, Ghatei MA, Bloom SR, Dhillo WS. The effects of kisspeptin-10 on reproductive hormone release show sexual dimorphism in humans. J Clin Endocrinol Metab. 2011 Dec;96(12):E1963-72. doi: 10.1210/jc.2011-1408. Epub 2011 Oct 5. PMID 21976724